CLINICAL TRIAL: NCT02516852
Title: Assessing the Effect of Sustainable Small-scale Egg Production on Maternal and Child Nutrition in Rural Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Community Markets for Conservation (COMACO) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1402004456
Record Dates: First submitted 2015-08-03; First posted 2015-08-06 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Malnutrition, Child; Malnutrition, Infant
Keywords: community development; poultry; animal-source food; stunting
MeSH Terms: conditions — Child Nutrition Disorders; Infant Nutrition Disorders; Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Egg production
- Control (No Intervention)

INTERVENTIONS:
Other: Egg production — Establishment and support of a community-owned and -operated egg production facility located at a central location in the community
  Arms: Intervention

SUMMARY:
Animal source foods (ASF), such as meat and eggs, are rich in nutrients critical for growth and development. Yet, for poor children in developing countries, ASF consumption is limited by cost, inadequate caregiver knowledge, and lack of local production and physical availability. The impact of HH- and village-level livestock interventions on household dietary diversity and nutritional status in resource-poor communities is not well established. The objective of this study is to test the effectiveness of local egg production intervention on maternal and child diets and child nutrition status.

This project takes place in the Luangwa Valley, Zambia in partnership with a local non-governmental organization, COMACO. Twenty communities will be assigned to the intervention, and 20 matched communities will be selected as controls. In each intervention community, an egg production facility will be built, owned, and operated by trained COMACO farmers.

Households (HHs) in each community will be sampled twice annually for 1 year pre-intervention (baseline) and 1 year post-intervention to assess dietary diversity and nutritional status. Data analysis will test for a change in these outcomes from baseline in each intervention community compared to the matched control community.

DETAILED DESCRIPTION:
The objective of this study is to test the effectiveness of an intervention establishing local egg production on maternal and child diets and nutrition status. The investigators hypothesize that this intervention, combined with appropriate agricultural extension and nutrition education programs, will result in: 1) increased total household, maternal, and child consumption of eggs; 2) improved maternal and child dietary quality; and 3) improved infant/ young child nutritional status.

The investigators will test this hypothesis in the Luangwa Valley, Zambia in partnership with a local non-governmental organization, Community Markets for Conservation (COMACO). The forty study sites are located in four geographic clusters (Chiefdoms) in Eastern Province Zambia. These Chiefdoms are located in two districts: Mambwe (Mnkhanya, Jumbe, and Nsefu Chiefdoms) and Lundazi (Mwanya Chiefdom).

Twenty communities will be assigned to the intervention (egg production), and 20 matched communities will be selected as controls (no intervention). In each intervention community, an egg production facility will be built, each owned and operated by trained COMACO farmers, mostly women. Each group will be provided layer pullets at point-of-lay and layer mash. Facility owners will make all business decisions, retain all profits, and will be responsible for all upkeep costs.

In a repeated cross-sectional study design, indicators of food security, wealth, diet, nutritional status (anthropometrics), and health and wellbeing will be assessed in all egg-producing HHs and in women/child dyads (children aged 6-36 months) residing in the area surrounding each facility or central control point. Data will be collected twice annually for 1 year pre-intervention (baseline) and 1 year post-intervention.

The exposure of interest is living in an egg-producing community. In the primary analysis, the investigators will use hierarchical mixed effects modeling to analyze the effect of the program on each of the outcomes of interest (see Outcome Measures section for details).

ELIGIBILITY:
Inclusion Criteria:

1. the HH dwelling is ≤1.5 km from the egg production facility or central control point;
2. there is a child 6-36 months of age in the HH; and,

Additionally, all HHs that include a member of the egg production group will be enrolled in the study, regardless of whether or not they meet the above inclusion criteria.

Exclusion Criteria:

1. the mother/primary caretaker or head of HH cannot converse with the field staff because of language;
2. the mother/primary caretaker or head of HH is unable to give informed consent or complete an interview without assistance; or,
3. the child is deformed, disabled, severely ill, or unable to cooperate for anthropometric measures.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3546 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in child height-for-age Z-score | 6, 12, 18, and 24 months after intervention
  Recumbent length for children < 24 months and standing height for those 24-36 months, with WHO Child Growth Standards as the reference population.

SECONDARY OUTCOMES:
Change in household egg consumption | 6, 12, 18, and 24 months after intervention
  7 day recall on total number of chicken or other eggs consumed in the household
Change in maternal egg consumption | 6, 12, 18, and 24 months after intervention
Change in child egg consumption | 6, 12, 18, and 24 months after intervention
Change in maternal dietary diversity | 6, 12, 18, and 24 months after intervention
  Measured by Women's Dietary Diversity Score, a 24 hour recall of all foods consumed, organized into 9 food groups
Change in child dietary diversity | 6, 12, 18, and 24 months after intervention
Change in child stunting | 6, 12, 18, and 24 months after intervention
  Defined as having a height-for-age z-score < -2.0, with WHO Growth Standards as the reference population.

OTHER OUTCOMES:
Change in household food security | 6, 12, 18, and 24 months after intervention
  Measure by Household Food Insecurity Access Scale (HFIAS), Household Hunger Scale (HHS) and/or Months of inadequate household food provisioning (MIHFP)
Change in producer household and poultry incomes | 6, 12, 18, and 24 months after intervention
Change in maternal physical and emotional health | 6, 12, 18, and 24 months after intervention
  Measured through a 6-item index adapted from RAND short form
Change in maternal nutritional status | 6, 12, 18, and 24 months after intervention
  Measured by mid-upper arm circumference and body mass index
Change in child weight-for-height Z-score | 6, 12, 18, and 24 months after intervention
Change in child weight-for-age Z-score | 6, 12, 18, and 24 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Travis, VMD, PhD, Principal Investigator — Cornell University
Locations (1):
- COMACO, Mfuwe, Eastern Province, Zambia

REFERENCES:
- See also: Community Markets for Conservation (COMACO) official website — http://www.itswild.org